CLINICAL TRIAL: NCT01873118
Title: READI (Readiness Evaluation And Discharge Interventions): Implementation as a Standard Nursing Practice for Hospital Discharge
Brief Title: READI (Readiness Evaluation And Discharge Interventions) Study
Acronym: READI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Marianne Weiss, Associate Professor, Marquette University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: ANCC2013-01
Record Dates: First submitted 2013-06-03; First posted 2013-06-07 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Discharge Transition of Patients Discharged to Home
Keywords: hospital discharge; discharge readiness; readmission; Emergency Department visits; Nurse assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Control hospital unit (No Intervention): This study involves implementation of interventions across entire hospital units. This arm is a usual care control unit paired to the intervention unit.
- implementation unit (Experimental): 3 implementation protocols implemented sequentially:
  1. RN-RHDS: implementation of discharge readiness assessment by the discharging nurse
  2. RN-RHDS+PT-RHDS: implementation of discharge readiness assessment by the discharging nurse which is informed by patient self-assessment of discharge readiness
  3. RN-RHDS+PT-RHDS+NIAF: implementation of discharge readiness assessment by the discharging nurse which is informed by patient self-assessment of discharge readiness followed by documentation of nurse actions initiated in response to the assessment. Nurse are instructed that action must be taken if any assessment item scores less than 7 ( on a 10 point scale).
  Interventions: Other: RN-RHDS protocol; Other: RN-RHDS+PT-RHDS protocol; Other: RN-RHDS + PT-RHDS + NIAF

INTERVENTIONS:
Other: RN-RHDS protocol — The discharging nurse assesses each patient being discharged home using the Readiness for Hospital Discharge Scale (RN version)
  Arms: implementation unit
Other: RN-RHDS+PT-RHDS protocol — The discharging nurse obtains and reviews patient self-report of discharge readiness using the Readiness for Hospital Discharge Scale - Patient version and then completes the Readiness for Hospital Discharge Scale (RN version)
  Arms: implementation unit
Other: RN-RHDS + PT-RHDS + NIAF — The discharging nurse assesses each patient being discharged home using the Readiness for Hospital Discharge Scale (RN version)after reviewing the patients self-perception of discharge readiness (PT-RHDS) and then records any actions taken in response to the discharge readiness assessment on the Nurse Initiated Action form (NIAF). When any item on the RN-RHDS is less than 7, an action is required.
  Arms: implementation unit

SUMMARY:
Preparation of patients for discharge is a primary function of hospital-based nursing care and readiness for discharge is an important outcome of hospital care. Inadequacies in discharge preparation have been well-documented and linked to difficulty with self-management after hospital discharge and with increased likelihood of emergency department (ED) use and readmission. Prior studies by the research team have led to recommendations for implementation of discharge readiness assessment as a standard nursing practice for hospital discharge.

The investigators will conduct a multi-site study to determine the impact on post-discharge utilization (readmission and ED visits) and costs of implementing discharge readiness assessment as a standard nursing practice for adult medical-surgical patients discharged to home. The study tests, in a stepped approach, the impact of implementing discharge readiness assessment by the discharging nurse as standard nursing practice (RN-RHDS protocol), the incremental value of informing the nurse assessment with the patient's perspective (RN-RHDS+PT-RHDS protocol), and of requiring that the nurse initiates and documents risk-mitigating actions for patients with low readiness scores (RN-RHDS+PT-RHDS+NIAF protocol).

HYPOTHESIS 1: Patients discharged using the RN-RHDS protocol will have fewer hospital readmissions and ED visits within 30 days post-discharge compared to patients discharged under usual care conditions.

HYPOTHESIS 2: Patients discharged using the RN-RHDS+PT-RHDS protocol will have fewer hospital readmissions and ED visits within 30 days post-discharge compared to patients discharged using the RN-RHDS protocol.

HYPOTHESIS 3: Patients discharged by nurses using the RN-RHDS+PT-RHDS protocol plus a Nurse-Initiated Action Form [NIAF] (RN-RHDS+PT-RHDS+NIAF protocol) will have fewer post-discharge readmissions and ED visits than patients discharged using the RN-RHDS+PT-RHDS protocol; the effect will be strongest for patients with low RHDS scores.

Aim 4: Conduct cost-benefit analysis of implementing discharge readiness assessment as standard practice, by comparing cost-savings from reduced post-discharge utilization against implementation costs.

ELIGIBILITY:
Inclusion Criteria:

* Medical, surgical, or medical-surgical nursing units of Magnet designated hospitals
* Patients 18 years of age or more, English speaking,able to read and understand consent who are being discharged to home as the discharge destination.
* Nursing personnel (Registered Nurses or Licensed Practical Nurses) who are performing discharge instructions and procedures on the day of hospital discharge.

Exclusion Criteria:

* Patients discharged to home with hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189796 (Actual)
Dates: Start 2014-07; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Post-discharge Utilization within 30 days after hospital discharge | 30 days after hospital discharge
  Readmissions and Emergency Department Visits within 30 days after hospital discharge

SECONDARY OUTCOMES:
Nurse Initiated Action Form | measured on day of hospital discharge typically 1 to 30 days after hospital admission
  Measures actions taken by the discharging nurse in response to discharge readiness assessment

OTHER OUTCOMES:
Readiness for Hospital Discharge Scale - RN version | measured on day of hospital discharge typically 1 to 30 days after hospital admission
  Nurses perceptions of patient readiness for hospital discharge
Readiness for Hospital Discharge Scale - Patient version | measured on day of hospital discharge typically 1 to 30 days after hospital admission
  Patient perception of discharge readiness

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Weiss, DNSc, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Bahr SJ, Bang J, Yakusheva O, Bobay KL, Krejci J, Costa L, Hughes RG, Hamilton M, Siclovan DM, Weiss ME. Nurse Continuity at Discharge and Return to Hospital. Nurs Res. 2020 May/Jun;69(3):186-196. doi: 10.1097/NNR.0000000000000417. PMID 31934945
- [Derived] Weiss ME, Yakusheva O, Bobay KL, Costa L, Hughes RG, Nuccio S, Hamilton M, Bahr S, Siclovan D, Bang J; READI Site Investigators. Effect of Implementing Discharge Readiness Assessment in Adult Medical-Surgical Units on 30-Day Return to Hospital: The READI Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e187387. doi: 10.1001/jamanetworkopen.2018.7387. PMID 30681712